CLINICAL TRIAL: NCT06580353
Title: Comparison of Viscoelastic Properties of Respiratory Muscles and Peripheral Muscles in Chronic Obstructive Pulmonary Disease Patients With Healthy Subjects
Brief Title: Viscoelastic Properties of Respiratory and Peripheral Muscles of COPD Patients
Status: Completed | Type: Observational
Sponsor: Gaziantep Islam Science and Technology University (Other)
Responsible Party: Principal Investigator, Çağtay Maden, Assistant professor, Gaziantep Islam Science and Technology University
Other Study IDs: 2023/391
Record Dates: First submitted 2024-08-26; First posted 2024-08-30 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-01

CONDITIONS: COPD; Muscle Tone Abnormalities
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COPD group: Patients with COPD who presented to the chest diseases polyclinic and whose symptoms of cough, sputum and/or dyspnoea accompanied by tachypnoea and/or tachycardia had not worsened in the last 14 days were defined as 'Stable COPD group' [
- Control group: The control group was defined as those who did not have any systemic disease and who were normal at the end of the polyclinic examination who applied to the chest diseases polyclinic.

SUMMARY:
The aim of this study was to compare the viscoelastic properties of auxiliary respiratory muscles and peripheral muscles of chronic obstructive pulmonary disease patients with healthy subjects. Myotonometry was used to evaluate the viscoelastic properties of the muscles. The viscoelastic properties of the sternoclaidus mastoid, pectoralis major, upper trapezius, deltoid, biceps brachii, rectus femoris, gastrocinemius, and tibialis anterior muscles were evaluated.

DETAILED DESCRIPTION:
muscle viscoelastic properties; muscle tone, stiffness and elasticity. These features may vary due to muscle overuse, lack of relaxation and recovery. The aim is to investigate these differences in COPD patients and healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* male gender,
* body mass index (BMI) between 18.5-29.9 kg/m2,
* stable COPD patients

Exclusion Criteria:

* being in the acute exacerbation period for COPD patients,
* having undergone any neurological, orthopaedic or thoracic surgery,
* presence of malignancy in any organ,
* presence of comorbidities affecting muscle atrophy (myasthenia gravis, muscular dystrophy, etc.).

Min Age: 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with COPD who visited the chest diseases clinic and had symptoms of cough, sputum, and/or shortness of breath, along with tachypnea and/or tachycardia, that had not worsened in the past 14 days were classified as the 'Stable COPD group'.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Respiratory functions (PEF) | 1 Day
  Peak expiratory flow (PEF) were measured was evaluated with spirometry. It will be recorded as liters and expected percentage
The Medical Research Council Scale | 1 Day
  Patients simply indicate on the scale the level of activity that causes dyspnoea in them according to the activities between 0-4.
The COPD Assessment Test | 1 Day
  This statement describes a scale consisting of eight items, each with response values ranging from 0 to 5. The total score is calculated by summing the responses to all the items, resulting in a range from 0 to 40. A higher total score indicates a greater negative impact of the disease on the individual's quality of life and daily activities.
Viscoelastic properties of muscles | 1 Day
  The viscoelastic properties of the muscles (muscle tone (Hz), and elasticity (Relative), stiffness (N/m)) were measured using a hand-held myotonometer.
Respiratory functions (FEV1) | 1 Day
  In pulmonary function test was evaluated with spirometry. forced expiratory volume in the first second (FEV1);will be recorded as liters and expected percentage
Respiratory functions (FVC) | 1 Day
  In pulmonary function test was evaluated with spirometry. forced expiratory volume in the first second (FEV1);will be recorded as liters and expected percentage
Respiratory functions (FEV1/FVC) | 1 Day
  ratio of forced expiratory volume in the first second to vital capacity (FEV1/FVC) was evaluated with spirometry.

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziantep İslamic Science and Technology University, Gaziantep, Şahinbey, Turkey (Türkiye)